CLINICAL TRIAL: NCT05248126
Title: Standard Patient Training Versus Vik Chatbot Guided Training: a Randomized Controlled Trial for Asthma Patients
Acronym: AsthmaTrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL21_0423 - UF7779; 2021-A02205-36 (Other: IDRCB number)
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Asthma
Keywords: chatbot; patient education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This prospective, randomized (1:1), controlled, pilot trial with a single-Zelen consent procedure will compare changes in quality of life, asthma control, lung function and health resource consumption between one group of patients with asthma participating in a classic treatment education program (the "standard education" arm) with a similar, second group of patients participating in a novel, chatbot-guided treatment education program (the "Vik" arm).
Masking Description: This protocol aims to compare two different ways of engaging with the patient and teaching. The notion of blinding per se is not adapted to this protocol, which is carried out, for all practical purposes, in an "open" fashion. Nevertheless, the Zelen randomisation procedure, which aims to maintain the comparator arm ignorant of the existence of the experimental arm in order to avoid "resentful demoralisation" effects, may also result in a partial blinding effect.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator arm (Active Comparator): All patients randomized to this arm will participate in a standard patient education program.
  Interventions: Other: Standard patient education
- Experimental arm (Experimental): All patients randomised to this arm have the opportunity to participate in a patient education programme via a chatbot.
  Interventions: Other: Chatbot patient education

INTERVENTIONS:
Other: Standard patient education — The comparator intervention is the usual therapeutic training for patients (ETP) cursus currently used in the General Pulmonology unit at the Arnaud De Villeneuve Hospital, Montpellier, France and approved by the French Regional Health Authority for the Occitanie Region [Agence Régional de Santé Occitanie].
  Arms: Comparator arm
Other: Chatbot patient education — The experimental intervention consists in providing the patient with access to a specific version of the "Vik-Asthme" chat bot for the duration of the study. Should the patient be unable to use or refuse to use the chatbot, the reasons for refusal will be documented and the patient will proceed with the comparator intervention.
  Arms: Experimental arm

SUMMARY:
The onset of smartphone usage has provided new opportunities for managing patients outside the walls of healthcare facilities. The development of asthma-specific smartphone applications represents an excellent area for partnership between developers and medical teams for delivering therapeutic education at the required time and in a personalised way. Within this context, the overall goal of the AsthmaTrain study is to perform a first, small pilot study comparing a new French-language chat-bot guided asthma patient education programme (the 'Vik' application) with the classic, authority-approved patient education program at the University Hospitals of Montpellier, Montpellier, France.

The primary objective is to compare a population of adult patients with asthma and participating in a standard patient education programme with a similar population participating in Vik-guided education programme in terms of change in overall scores on the Asthma Quality of Life Questionnaire (AQLQ).

DETAILED DESCRIPTION:
Secondarily, the following will also be compared between the two study arms:

* the subdomains of the AQLQ score,
* lung function, overall asthma control and exacerbation rates,
* general health status via the Euroqol 5-domain 5-level questionnaire (EQ-5D-5L),
* adherence to the program and burden of the program for the medical team,
* major categories of direct health resource consumption.

Finally, because education intervention success may depend on patient-specific characteristics, an ancillary study will compare the following baseline traits between the 50% best intervention responders in either arm:

* the big five personality traits,
* the hospital anxiety and depression,
* coping mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 18
* Physician-confirmed diagnosis of asthma

Exclusion Criteria:

* Protected populations according to the French Public Health Code Articles L1121-6,8
* The subject has already participated in the present study
* Subject unable to comply with trial procedures/visits
* Potential for interference from another study
* Non-beneficiary of the French single-payer national medical insurance system
* Lack of informed consent
* Patients already using the Vik Asthma application in their daily lives or having already followed a therapeutic education program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Change in the total AQLQ score | baseline to 6 months
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain instrument that can either be self- or interviewer-administered. The recall-time is two weeks. The four domains covered are: (i) symptoms (11 items), (ii) activity limitation (12 items, 5 of which are individualized), (iii) emotional function (5 items), and (iv) environmental exposure (4 items). Each item is ranked by the patient using a 7-point Likert scale ranging from 1 (severely impaired) to 7 (not impaired at all). Scores range from 1 to 7, higher scores indicate better quality of life and a minimally important difference (for overall scores and for each sub-domain) has been established at 0.5.

SECONDARY OUTCOMES:
Change in the 'symptoms' domain of the AQLQ from baseline to six months | baseline to 6 months
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain instrument that can either be self- or interviewer-administered. The recall-time is two weeks. The four domains covered are: (i) symptoms (11 items), (ii) activity limitation (12 items, 5 of which are individualized), (iii) emotional function (5 items), and (iv) environmental exposure (4 items). Each item is ranked by the patient using a 7-point Likert scale ranging from 1 (severely impaired) to 7 (not impaired at all). Scores range from 1 to 7, higher scores indicate better quality of life and a minimally important difference (for overall scores and for each sub-domain) has been established at 0.5.
Change in the 'activity limitation' domain of the AQLQ from baseline to six months | baseline to 6 months
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain instrument that can either be self- or interviewer-administered. The recall-time is two weeks. The four domains covered are: (i) symptoms (11 items), (ii) activity limitation (12 items, 5 of which are individualized), (iii) emotional function (5 items), and (iv) environmental exposure (4 items). Each item is ranked by the patient using a 7-point Likert scale ranging from 1 (severely impaired) to 7 (not impaired at all). Scores range from 1 to 7, higher scores indicate better quality of life and a minimally important difference (for overall scores and for each sub-domain) has been established at 0.5.
Change in the 'emotional function' domain of the AQLQ from baseline to six months | baseline to 6 months
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain instrument that can either be self- or interviewer-administered. The recall-time is two weeks. The four domains covered are: (i) symptoms (11 items), (ii) activity limitation (12 items, 5 of which are individualized), (iii) emotional function (5 items), and (iv) environmental exposure (4 items). Each item is ranked by the patient using a 7-point Likert scale ranging from 1 (severely impaired) to 7 (not impaired at all). Scores range from 1 to 7, higher scores indicate better quality of life and a minimally important difference (for overall scores and for each sub-domain) has been established at 0.5.
Change in the 'environmental exposure' domain of the AQLQ from baseline to six months | baseline to 6 months
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain instrument that can either be self- or interviewer-administered. The recall-time is two weeks. The four domains covered are: (i) symptoms (11 items), (ii) activity limitation (12 items, 5 of which are individualized), (iii) emotional function (5 items), and (iv) environmental exposure (4 items). Each item is ranked by the patient using a 7-point Likert scale ranging from 1 (severely impaired) to 7 (not impaired at all). Scores range from 1 to 7, higher scores indicate better quality of life and a minimally important difference (for overall scores and for each sub-domain) has been established at 0.5.
Change in the ACQ-5 score | baseline to 6 months
  The ACQ-5 is a shortened version of the ACQ that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) omitting the forced expiratory volume in 1 second measurement and short acting beta antagonist use from the original ACQ score. Patients are asked to recall how their asthma has been during the previous week by responding to 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-5 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma . Individual changes of at least 0.5 are considered to be clinically meaningful.
Change in %predicted values of forced expiratory volume in 1 second (FEV1) | baseline to 6 months
Change in %predicted values of forced vital capacity (FVC) | baseline to 6 months
Change in FEV1/FVC ratios (litres/litres) | baseline to 6 months
Change in the EQ-5D-5L score | baseline to 6 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Percentage of patients participating in the 6 month visit | 6 months
For the experimental arm only, weeks of chatbot usage | baseline to 6 months
Cumulative number of emails to/from the patient | baseline to 6 months
Cumulative number of telephone calls to/from the patient | baseline to 6 months
The cumulative dose for short-acting beta antagonists | baseline to 6 months
The cumulative dose for long acting beta antagonists | baseline to 6 months
The cumulative dose for short acting muscarinic antagonists | baseline to 6 months
The cumulative dose for long acting muscarinic antagonists | baseline to 6 months
The cumulative dose for oral corticosteroids | baseline to 6 months
The cumulative dose for inhaled corticosteroids | baseline to 6 months
The cumulative dose for nasal corticosteroids | baseline to 6 months
Accumulating numbers of generalist consults | baseline to 6 months
Accumulating numbers of specialist consults | baseline to 6 months
Accumulating numbers of nursing consults | baseline to 6 months
Accumulating numbers of unexpected/emergency consults | baseline to 6 months
Accumulating numbers of days of hospitalization (in relation to asthma) | baseline to 6 months
Accumulating numbers of days of intensive care (in relation to asthma) | baseline to 6 months
Accumulating numbers of days of exacerbation | baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study.
  Data will be made available to persons who address a reasonable request to the study director.
  Individual participant data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  The study protocol, participant information materials, and paper case report form will also be made available to the public.
Supporting Information: Study Protocol
Time Frame: Datasets that underlie the results reported in the article (text, tables, figures, and appendices) can be requested after the publication process has been completed.
  The protocol will be published in an open-access journal. The remaining documents will be made available on the Open Science Framework as they are finalized.
Access Criteria: * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
  * If the data do not fulfil the requirements of the reference methodology (MR-001) (ex: data about religion, etc.), the appropriate CNIL (National Commission for Computing and Liberties) approval has to be obtained by the user.
  * If the data will be used outside the European Union, standard contractual clauses have to be signed between Montpellier University Hospital and the user before sharing data.
URL: https://osf.io/u972h/

REFERENCES:
- [Background] Suehs CM, Vachier I, Galeazzi D, Vaast F, Cardon F, Molinari N, Bourdin A. Standard patient training versus Vik-Asthme chatbot-guided training: 'AsthmaTrain' - a protocol for a randomised controlled trial for patients with asthma. BMJ Open. 2023 Feb 21;13(2):e067039. doi: 10.1136/bmjopen-2022-067039. PMID 36810168